CLINICAL TRIAL: NCT04011475
Title: Taiwan Outcomes and Real-world Treatment Options for Chronic Obstructive Pulmonary Disease
Brief Title: A Study in Taiwan Based on Medical Records That Looks at the Occurrence of Flare-ups in Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Started LABA/LAMA or LAMA Treatment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0086
Record Dates: First submitted 2019-06-28; First posted 2019-07-08 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subjects with Tiotropium and Olodaterol
  Interventions: Drug: Tiotropium + Olodaterol
- Subjects treated with other LABA/LAMA therapy
  Interventions: Drug: Other LABA/LAMA
- Subjects treated with LAMA therapy
  Interventions: Drug: LAMA

INTERVENTIONS:
Drug: Tiotropium + Olodaterol — Spiolto®
  Groups: Subjects with Tiotropium and Olodaterol
Drug: Other LABA/LAMA — tiotropium/olodaterol, indacaterol/glycopyrronium, vilanterol/umeclidinium
  Groups: Subjects treated with other LABA/LAMA therapy
Drug: LAMA — aclidinium bromide, glycopyrronium, tiotropium, umeclidinium
  Groups: Subjects treated with LAMA therapy

SUMMARY:
Study to collect the data on Chronic Obstructive Pulmonary Disease (COPD) patients who were administered with Long-Acting Beta-Agonist/ Long-Acting Muscarinic Antagonist (LABA/LAMA) (Fixed-dose Combination (FDC) or free combo) or LAMA treatment

ELIGIBILITY:
Inclusion Criteria:

Patients who fulfil ALL the following criteria are included.

1. Patients who diagnosed with COPD who were prescribed with LABA/LABA (FDC or free combo) as a new initiation or switching from other therapy (i.e., single/dual/triple), or newly receiving LAMA treatment for 3 months at least prior to 30 June 2018
2. Male or female patients ≥ 40 years of age

Exclusion Criteria:

1. Patients who meet the following criterion are not included.

* Patients with documented diagnosis of bronchial asthma, asthma-COPD overlap syndrome (ACOS), bronchiectasis, cystic fibrosis, or lung cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data will be retrospectively abstracted from the medical chart after eligibility assessment. Eligible patients will be categorized into the cohort A (patients treated with Tio + Olo), B (patients treated with other LABA/LAMA therapy), and C (patients treated with LAMA therapy).
Sampling Method: Non-Probability Sample
Enrollment: 1617 (Actual)
Dates: Start 2019-12-29 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Taiwan (12):
  - Ditmanson Medical Foundation Chia - Yi Christian Hospital, Chia YI City
  - CGMH Chia YI, Chia YI City
  - Eda hospital, Kaohsiung City
  - CGMH Kaohsiung, Kaohsiung City
  - Far east memorial hospital, New Taipei City
  - China medicine memorial hospital, Taichung
  - VGH Taichung, Taichung
  - National Taiwan University hospital, Taipei
  - Makay memorial hospital, Taipei
  - Cheng Hsin general hospital, Taipei
  - Taipei Tzu Chi hospital, Taipei
  - CGMH Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective, multi-center, cohort study to collect the data on Chronic Obstructive Pulmonary Disease (COPD) patients in Taiwan who were administered with tiotropium + olodaterol, other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Fixed-dose Combination (FDC) or free combo) or LAMA treatment for 3 months investigating the occurrence of COPD exacerbations among such patients.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Only subjects who strictly met all inclusion and none of the exclusion criteria were included in the study.
Groups:
- Tiotropium+Olodaterol (Group A): Eligible Chronic Obstructive Pulmonary Disease (COPD) patients in Taiwan who were administered with tiotropium + olodaterol for 3 months at least prior to 30 June 2018 were included in this group.
- Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B): Eligible Chronic Obstructive Pulmonary Disease (COPD) patients in Taiwan who were administered with other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (fixed-dose combinations (FDC)/free combos) for 3 months at least prior to 30 June 2018 were included in this group.
- Long-Acting Muscarinic Antagonist (LAMA) (Group C): Eligible Chronic Obstructive Pulmonary Disease (COPD) patients in Taiwan who were administered with other Long-Acting Muscarinic Antagonist (LAMA) for 3 months at least prior to 30 June 2018 were included in this group.
Period: Overall Study
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Started | 239 | 937 | 441
Propensity Score Matched Cohort (Eligible patients matching via propensity score to balance the baseline characteristics between study groups.) | 114 | 114 | 114
Completed | 239 | 937 | 441
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score matched cohort: All eligible Chronic Obstructive Pulmonary Disease (COPD) patients in Taiwan who were administered with tiotropium + olodaterol, other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Fixed-dose Combination (FDC) or free combo) or LAMA treatment for 3 months at least prior to 30 June 2018, and matching via propensity score to balance the baseline characteristics between the study groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C) | Total
Number analyzed (Participants) | 114 | 114 | 114 | 342
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (9.99) | 71.6 (9.54) | 71.0 (9.37) | 71.3 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 24
  Male | 106 | 106 | 106 | 318
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 114 | 114 | 114 | 342
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate-to-severe Acute Exacerbation
Description: Number of participants with moderate-to-severe acute exacerbation within 1 year after the index date was reported.
Time Frame: Up to 1 year after the index date (Baseline).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
Participants | 20 | 22 | 9
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0276, Log Rank
Statistical Analysis 2: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.6665, Regression, Cox; Hazard Ratio (HR) = 0.875, 95% CI 2-sided [0.47 to 1.604] — Hazard Ratio (HR) was from Cox regression comparing group A versus group B using group B as reference
Statistical Analysis 3: Comparison: Tiotropium+Olodaterol (Group A) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0310, Regression, Cox; Hazard Ratio (HR) = 2.377, 95% CI 2-sided [1.083 to 5.221] — Hazard Ratio (HR) was from Cox regression comparing group A versus group C using group C as reference
Statistical Analysis 4: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0116, Regression, Cox; Hazard Ratio (HR) = 2.716, 95% CI 2-sided [1.250 to 5.901] — Hazard Ratio (HR) was from Cox regression comparing group B versus group C using group C as reference

2. Secondary Outcome: Annualized Rate of Moderate-to-severe Exacerbation
Description: The annualized rate of moderate-to-severe exacerbation was calculated as: total number of episodes of moderate-to-severe exacerbation of all participants divided by the sum of follow-up period [years] of all participants. The corresponding 95% confidence interval was from Poisson regression.
Time Frame: Up to 1 year after the index date (Baseline).
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: episodes/patient-year
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
episodes/patient-year | 0.28 [0.20 to 0.40] | 0.42 [0.32 to 0.56] | 0.10 [0.05 to 0.17]
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.0756, Z-test; Rate ratio = 0.67, 95% CI 2-sided [0.43 to 1.04] — The rate ratio was from Poisson regression for Group A versus Group B using Group B as the reference group
Statistical Analysis 2: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p < 0.0001, Z-test; Rate ratio = 4.36, 95% CI 2-sided [2.27 to 8.40] — The rate ratio was from Poisson regression for Group B versus Group C using Group C as the reference group
Statistical Analysis 3: Comparison: Tiotropium+Olodaterol (Group A) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0022, Z-test; Rate ratio = 0.34, 95% CI 2-sided [0.17 to 0.68] — The rate ratio was from Poisson regression for Group C versus Group A using Group A as the reference group

3. Secondary Outcome: Annualized Rate of Mild Exacerbation
Description: The annualized rate of mild exacerbation was calculated as: total number of episodes of mild exacerbation of all participants divided by the sum of follow-up period [years] of all participants. The corresponding 95% confidence interval was from Poisson regression.
Time Frame: Up to 1 year after the index date (Baseline).
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: episodes/patient-year
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
episodes/patient-year | 0.00 [0.00 to NA] — Since no subject experienced mild acute exacerbation during this period, the upper limit of the rate was divergent to infinity and hence, not available. | 0.04 [0.02 to 0.11] | 0.04 [0.01 to 0.09]
Statistical Analysis 1: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.7394, Z-test; Rate ratio = 1.25, 95% CI 2-sided [0.34 to 4.65] — The rate ratio was from Poisson regression for Group B versus Group C using Group C as the reference group

4. Secondary Outcome: Annualized Rate of Moderate Exacerbation
Description: The annualized rate of moderate exacerbation was calculated as: total number of episodes of moderate exacerbation of all participants divided by the sum of follow-up period [years] of all participants. The corresponding 95% confidence interval was from Poisson regression.
Time Frame: Up to 1 year after the index date (Baseline).
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: episodes/patient-year
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
episodes/patient-year | 0.19 [0.13 to 0.29] | 0.30 [0.21 to 0.42] | 0.08 [0.04 to 0.15]
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.1116, Z-test; Rate ratio = 0.65, 95% CI 2-sided [0.38 to 1.11] — The rate ratio was from Poisson regression for Group A versus Group B using Group B as the reference group
Statistical Analysis 2: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0004, Z-test; Rate ratio = 3.78, 95% CI 2-sided [1.81 to 7.88] — The rate ratio was from Poisson regression for Group B versus Group C using Group C as the reference group
Statistical Analysis 3: Comparison: Tiotropium+Olodaterol (Group A) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0239, Z-test; Rate ratio = 0.41, 95% CI 2-sided [0.19 to 0.89] — The rate ratio was from Poisson regression for Group C versus Group A using Group A as the reference group

5. Secondary Outcome: Annualized Rate of Severe Exacerbation
Description: The annualized rate of severe exacerbation was calculated as: total number of episodes of severe exacerbation of all participants divided by the sum of follow-up period [years] of all participants. The corresponding 95% confidence interval was from Poisson regression.
Time Frame: Up to 1 year after the index date (Baseline).
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: episodes/patient-year
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
episodes/patient-year | 0.09 [0.05 to 0.16] | 0.12 [0.07 to 0.21] | 0.02 [0.00 to 0.07]
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.4164, Z-test; Rate ratio = 0.71, 95% CI 2-sided [0.32 to 1.61] — The rate ratio was from Poisson regression for Group A versus Group B using Group B as the reference group
Statistical Analysis 2: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0100, Z-test; Rate ratio = 7.00, 95% CI 2-sided [1.59 to 30.8] — The rate ratio was from Poisson regression for Group B versus Group C using Group C as the reference group
Statistical Analysis 3: Comparison: Tiotropium+Olodaterol (Group A) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0377, Z-test; Rate ratio = 0.20, 95% CI 2-sided [0.04 to 0.91] — The rate ratio was from Poisson regression for Group C versus Group A using Group A as the reference group

6. Secondary Outcome: Incidence of Patients Escalating Therapy (From Single/Dual to Dual/Triple Therapy)
Description: Incidence of patients escalating therapy, from single/dual to dual/triple therapy such as receiving Long-Acting Muscarinic Antagonist (LAMA) escalated to dual therapy or receiving LABA+LAMA (Tiotropium+Olodaterol) escalated to triple therapy(LABA+LAMA+inhaled corticosteroids (ICS)), within 1 year after the index date was reported.
Time Frame: Up to 1 year after the index date (Baseline).
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
Participants | 10 | 17 | 19
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.2035, Log Rank

7. Secondary Outcome: Percentage of Patients Receiving Dual Therapy Escalated to Triple Therapy or LAMA Escalated to Dual Therapy
Description: Percentage of patients receiving dual therapy (Tiotropium+Olodaterol or other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) therapy) escalated to triple therapy (LABA+LAMA + inhaled corticosteroids (ICS)) or LAMA escalated to dual therapy (LABA + LAMA) was reported.
Time Frame: Up to 1 year after index date (Baseline).
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
Percentage of participants | 8.8 | 14.9 | 16.7
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.1858, Chi-squared; Chi-square test was applied for assessing the inter-group difference

8. Secondary Outcome: Change From Baseline in Pulmonary Function After LABA+LAMA or LAMA Initiation Evaluating by Post-bronchodilator Forced Expiratory Volume in One Second (Post-FEV1) at 12 Months After Index Date
Description: Change from baseline in pulmonary function after Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Tiotropium+Olodaterol or other LABA+LAMA therapy) or LAMA initiation evaluating by post-bronchodilatorForced Expiratory Volume in one second (Post-FEV1) at 12 months after index date was reported.
  Spirometry was the most common tool to evaluate the lung function of patients with respiratory disease. Among the results of spirometry, post-bronchodilator Forced Expiratory Volume in one second was used for assisting in the diagnosis, determining disease severity, and following up the prognosis.
Time Frame: At index date (Baseline) and at 12 months after index date.
Population: Propensity score (PS) matched cohort: All eligible Chronic Obstructive Pulmonary Disease patients in Taiwan who were administered with tiotropium + olodaterol, other Long-Acting Beta-Agonist +Long-Acting Muscarinic Antagonist (LAMA) (Fixed-dose Combination or free combo) or LAMA treatment for 3 months at least prior to 30 June 2018, and matching via PS to balance the baseline characteristics between the study groups. Only patients with non-missing endpoint results were included in the analysis.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 15 | 11 | 19
milliliter | -142.0 (197.02) | 20.0 (240.46) | -2.1 (176.05)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A); Test type: Other; p = 0.0144, Pair t-test; Pair t-test was used for assessing the intra-group difference
Statistical Analysis 2: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.9219, Pair t-test; Pair t-test was used for assessing the intra-group difference
Statistical Analysis 3: Comparison: Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.9590, Pair t-test; Pair t-test was used for assessing the intra-group difference

9. Secondary Outcome: Change From Baseline in Pulmonary Function After LABA+LAMA or LAMA Initiation Evaluating by Post-bronchodilator Forced Volume Vital Capacity (Post-FVC) at 12 Months After Index Date
Description: Change from baseline in pulmonary function after Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Tiotropium+Olodaterol or other LABA+LAMA therapy) or LAMA initiation evaluating by post-bronchodilator Forced Volume Vital Capacity (Post-FVC) at 12 months after index date was reported.
  Spirometry was the most common tool to evaluate the lung function of patients with respiratory disease. Among the results of spirometry, post-bronchodilator Forced Volume Vital Capacity was used for assisting in the diagnosis, determining disease severity, and following up the prognosis.
Time Frame: At index date (Baseline) and at 12 months after index date.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 15 | 11 | 19
milliliter | -74.0 (261.09) | 134.5 (295.38) | 63.7 (375.67)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A); Test type: Other; p = 0.2909, Pair t-test; Pair t-test was used for assessing the intra-group difference
Statistical Analysis 2: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.1618, Pair t-test; Pair t-test was used for assessing the intra-group difference
Statistical Analysis 3: Comparison: Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.4695, Pair t-test; Pair t-test was used for assessing the intra-group difference

10. Secondary Outcome: Change From Baseline in Pulmonary Function After LABA+LAMA or LAMA Initiation Evaluating by COPD Assessment Test (CAT) Score at 12 Months After Index Date
Description: Change from baseline in pulmonary function after Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Tiotropium+Olodaterol or other LABA+LAMA therapy) or LAMA initiation evaluating by Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) score at 12 months after index date was reported.
  The COPD assessment test (CAT) was a simple, 8-item, health status instrument which provided a simple method for assessing the impact of COPD on the patient's health and the quality of life. Each item was on a 6-point scale: 0 (no impact) to 5 (maximum impact). The CAT score ranging from 0 (better health status) to 40 (worse health status) was calculated by summing the points for each item. A decrease in CAT score represents an improvement in health status, whereas an increase in CAT score represents a worsening in health status.
Time Frame: At index date (Baseline) and at 12 months after index date.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 31 | 26 | 31
Score on a scale | 0.0 (5.40) | 1.0 (4.51) | 2.4 (5.05)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A); Test type: Other; p > 0.9999, Pair t-test; Pair t-test was used for assessing the intra-group difference
Statistical Analysis 2: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.2516, Pair t-test; Pair t-test was used for assessing the intra-group difference
Statistical Analysis 3: Comparison: Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0036, Pair t-test; Pair t-test was used for assessing the intra-group difference

11. Secondary Outcome: Change From Baseline in Pulmonary Function After LABA+LAMA or LAMA Initiation Evaluating by Modified Medical Research Council Dyspnea Scale (mMRC) at 12 Months After Index Date
Description: Change from baseline in pulmonary function after Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Tiotropium+Olodaterol or other LABA+LAMA therapy) or LAMA initiation evaluating by modified Medical Research Council dyspnea scale (mMRC) at 12 months after index date is reported.
  Modified Medical Research Council dyspnea scale (mMRC) is a 5 points scale measuring the severity of dyspnea of patients. The scale ranges from 0 (better outcome) to 4 (worse outcome). The higher the scale value, the more severe the dyspnea is. If mMRC scale of the patient was > 2, it means the patient may suffer from dyspnea.
Time Frame: At index date (baseline) and at 12 months after index date
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 28 | 23 | 21
Score on a scale | 0.1 (1.07) | 0.1 (0.67) | 0.2 (0.68)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A); Test type: Other; p = 0.6189, Wilcoxon (Mann-Whitney); Wilcoxon test was used for assessing the intra-group difference
Statistical Analysis 2: Comparison: Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B); Test type: Other; p = 0.7656, Wilcoxon (Mann-Whitney); Wilcoxon test was used for assessing the intra-group difference
Statistical Analysis 3: Comparison: Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.3594, Wilcoxon (Mann-Whitney); Wilcoxon test was used for assessing the intra-group difference

12. Secondary Outcome: Percentage of Patients Using Rescue Medications
Description: Percentage of patients using rescue medications within 1 year after index date was reported.
Time Frame: Up to 1 year after index date (Baseline).
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
Number analyzed (Participants) | 114 | 114 | 114
Percentage of participants | 58.8 | 43.9 | 45.6
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (Group A) vs Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) vs Long-Acting Muscarinic Antagonist (LAMA) (Group C); Test type: Other; p = 0.0483, Chi-squared; Chi-square test was applied for assessing the inter-group difference

ADVERSE EVENTS:
Time Frame: Up to 1 year after the index date (Baseline).
Description: All eligible Chronic Obstructive Pulmonary Disease (COPD) patients in Taiwan who were administered with tiotropium + olodaterol, other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Fixed-dose Combination (FDC) or free combo) or LAMA treatment for 3 months at least prior to 30 June 2018. Only adverse drug reactions and adverse events with fatal outcomes were collected.
Arm/Group | Tiotropium+Olodaterol (Group A) | Other Long-Acting Beta-Agonist (LABA)+Long-Acting Muscarinic Antagonist (LAMA) (Group B) | Long-Acting Muscarinic Antagonist (LAMA) (Group C)
All-Cause Mortality (participants affected / at risk) | 0/239 | 0/937 | 0/441
Serious Adverse Events (participants affected / at risk) | 0/239 | 0/937 | 0/441
Other Adverse Events (participants affected / at risk) | 0/239 | 0/937 | 0/441

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT04011475/Prot_SAP_000.pdf